CLINICAL TRIAL: NCT05640921
Title: Group-integrated Cognitive Behavioural Therapy (Gi-CBT) to Aid Communities' Reintegration of Former Terrorists in Nigeria: A Randomised Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Teesside University (Other)
Collaborators: Coal City University (Unknown)
Responsible Party: Principal Investigator, Tarela Ike, Dr, Teesside University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0000-0003-0516-0313c
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Depression; Trauma; Anxiety; Fear
MeSH Terms: conditions — Depression; Wounds and Injuries; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-integrated Cognitive Behavioural Therapy (Gi-CBT) (Experimental): The Gi-CBT sessions will cover relevant aspects of tackling trauma, and the CBT component will involve addressing negative thoughts, building more positive ones and building resilience through post-traumatic situations and adversities.
  Interventions: Behavioral: Gi-CBT
- Media Intervention (Active Comparator): The second group will receive Media Orientation (MO). The MO sessions will embed media content to create awareness of the government's approaches to reintegration.
  Interventions: Other: Media Orientation

INTERVENTIONS:
Behavioral: Gi-CBT — Gi-CBT designed to cover relevant aspects of tackling trauma, and the CBT component will involve addressing negative thoughts, building more positive ones and building resilience.
  Arms: Group-integrated Cognitive Behavioural Therapy (Gi-CBT)
Other: Media Orientation — The MO sessions will embed media content to create awareness of the government's approaches to reintegration.
  Arms: Media Intervention

SUMMARY:
The project aims to make significant contributions that change the conversation in communities and policy circles through promoting knowledge of nonviolent peace strategies using the Group integrated Cognitive Behavioural Therapy (Gi-CBT) to help heal trauma, improve peace, and encourage positive rehabilitation and reintegration of former Boko Haram terrorists' members and their families.

DETAILED DESCRIPTION:
The main question it aims to answer are:

• What is the feasibility in terms of recruitment, retention, adherence to the intervention and communities/victims' satisfaction with Gi-CBT to promote healing and improve the successful reintegration of of former Boko Haram terrorists' members and their families.into society?

Participants will be randomly allocated into two groups. The first group, the intervention group, will receive the Group integrated Cognitive Behavioural Therapy (Gi-CBT). The second group will receive government intervention involving media messages from the National Orientation Agency devoid of GiCBT.

Researchers will compare Gi-CBT group with the media orientation group to see if there are differences between a change in attitude towards ex-offenders' reintegration at base line, end of intervention and three months follow up.

ELIGIBILITY:
Inclusion Criteria:

1. community members who had previous experience of trauma as a result of Boko Haram atrocities, score 5 and above for the culturally-adapted Trauma Screening Questionnaire (Brewinn et al., 2002)
2. are aged 18+ years and above
3. are residents of the designated areas including Bornu (Maiduguri), and its environs.

Exclusion Criteria:

* those not meeting the study inclusion criteria will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Service Satisfaction Scale | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months post-intervention]
  Change in service satisfaction is being assessed
PHQ-9 | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months post-intervention]
  Change in Depressive Symptoms
The Attitude Towards Repentant Terrorist and their Reintegration scale | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months post-intervention]
  Change in attitude towards reintegration
Trauma Screening Questionnaire | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months post-intervention
  Change in traumatic experience is being assessed

IPD SHARING:
Plan to Share IPD: No